CLINICAL TRIAL: NCT07225855
Title: Geriatric Assessment and Management for Older Adults Undergoing Radiation Therapy for Head and Neck Cancer and Their Family Caregivers
Brief Title: Geriatric Assessment and Management for Older Adults Undergoing Chemotherapy and Radiation Therapy for Head and Neck Cancer and Their Family Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22617; NCI-2025-07662 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22617 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Localized Head and Neck Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Health Communication; Interviews as Topic; Office Visits; Referral and Consultation; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (GA-driven intervention) (Experimental): Patients undergo PGA at baseline, at 4 weeks and at 1 month after completing treatment. Assessment results shared with treating oncologists and patients receive referrals to supportive care services for the problems identified with the assessment throughout the study. Caregivers may receive referrals to resources and programs.
  Interventions: Other: Electronic Health Record Review; Behavioral: Health Communication; Other: Interview; Other: Practical Geriatric Assessment; Other: Questionnaire Administration; Other: Referral; Other: Supportive Care
- Arm B (usual care) (Active Comparator): Patients attend regular clinical visits for treatment and follow up and receive usual care provided by their radiation oncology and medical oncology teams and referrals to supportive care services as needed throughout the study.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review; Other: Office Visit; Other: Questionnaire Administration; Other: Referral

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm B (usual care)
Other: Electronic Health Record Review — Ancillary studies
Behavioral: Health Communication — Shared with treating oncology
  Arms: Arm A (GA-driven intervention)
Other: Interview — Ancillary studies
  Arms: Arm A (GA-driven intervention)
Other: Office Visit — Attend regular clinical visits
  Arms: Arm B (usual care)
Other: Practical Geriatric Assessment — Undergo PGA
  Arms: Arm A (GA-driven intervention)
Other: Questionnaire Administration — Ancillary studies
Other: Referral — Receive referrals to resources and programs
  Other Names: Referred
  Arms: Arm A (GA-driven intervention)
Other: Referral — Receive referrals to supportive care services
  Other Names: Referred
  Arms: Arm B (usual care)
Other: Supportive Care — Receive referrals to supportive care services
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Arm A (GA-driven intervention)

SUMMARY:
This clinical trial compares the effect of geriatric assessment (GA)-based management of supportive care to usual care in treating older patients undergoing chemotherapy and radiation therapy for head and neck cancer and their family caregivers (FCG). At least one quarter of head and neck cancers patients are diagnosed at age 70 or older. Treatment for head and neck cancers usually include surgery, chemotherapy, and radiation. Older adults are often at higher risk for functional problems, and may experience more side effects. In addition, there may be a lack of support mechanisms in place to address the needs of these older patients. Cancer not only affects the patients but the entire family, especially the family member who is the caregiver. Currently, all patients over 65 receive the same standard of care based on national guidelines, which include supportive care referrals. However, data suggests, that many patients may need more frequent and structured support. The Practical Geriatric Assessment (PGA) is a complete examination including evaluation of the physical and mental function as well as the emotional state of the older patient. PGA-based supportive care interventions may be safe, tolerable, and/or effective in managing treatment-related side effects and improving quality of life compared to usual care in older patients undergoing chemotherapy and radiation therapy for head and neck cancer and their FCG.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of the intervention by evaluation of treatment-related toxicities.

SECONDARY OBJECTIVES:

I. To assess the feasibility, retention, and acceptability of the intervention. II. To assess the rate of any grade non-hematologic treatment-related toxicities.

III. To assess patient/FCG self-reported outcomes. IV. To assess the symptom-related outcomes by evaluation of unplanned readmissions and emergency room (ER)/urgent care visits.

OUTLINE: Patients are randomized to 1 of 2 arms. Caregivers are randomized to the same arm as the corresponding patients.

ARM A (GA-DRIVEN INTERVENTION): Patients undergo PGA at baseline, at 4 weeks and at 1 month after completing treatment. Assessment results shared with treating oncologists and patients receive referrals to supportive care services for the problems identified with the assessment throughout the study. Caregivers may receive referrals to resources and programs.

ARM B (USUAL CARE): Patients attend regular clinical visits for treatment and follow up and receive usual care provided by their radiation oncology and medical oncology teams and referrals to supportive care services as needed throughout the study.

After completion of study interventions, patients are followed up at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Documented written informed consent of the participant
* PATIENT: Diagnosis of non-metastatic head and neck cancer
* PATIENT: Age: ≥ 60 years
* PATIENT: Patient must be scheduled to undergo curative-intent, definitive radiation with or without concurrent chemotherapy or postoperative radiation with or without concurrent chemotherapy
* PATIENT: Patients must have at least one geriatric assessment as assessed by the modified Geriatric 8 (G8) tool
* PATIENT: Family caregivers (FCGs) are highly encouraged to participate but this is not required. Patients without FCGs will be eligible to participate in the study. FCGs will be randomized to the same arm as their corresponding patients
* PATIENT: Ability to read and understand English
* CAREGIVER: A family member or friend identified by the patient and defined as a person who knows the patient well and is involved in the patient's medical care
* CAREGIVER: Ability to read and understand English
* CAREGIVER: Age 18 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-07-09 (Estimated); Primary Completion 2027-11-24 (Estimated); Study Completion 2027-11-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of grade 2-5 non-hematologic treatment-related toxicities | Up to 3 months after completion of treatment
  Will be assessed in patients using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Will be summarized using descriptive statistics. For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Observed toxicities will be summarized by type, severity, and attribution. Rates will be estimated along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Percentage of eligible participants who enroll in the study | Up to 1 year
  The denominator will be all patients who meet eligibility criteria and are approached for consent. The numerator will be those who provide consent and are successfully randomized. The feasibility threshold will be met if ≥ 60% of eligible patients enroll and are randomized. Will be summarized using descriptive statistics. Rates will be estimated along with the 95% exact binomial confidence interval.
Retention rate | Up to 3 months after completion of study treatment
  Will be defined as the percentage of participants in the intervention arm who complete the Practical Geriatric Assessment (PGA) tool. The denominator will be all patients randomized to the intervention arm. The retention threshold will be met if ≥ 60% of these participants complete the PGA tool. Will be summarized using descriptive statistics. Rates will be estimated along with the 95% exact binomial confidence interval.
Acceptability of the intervention | Up to 3 months after completion of treatment
  Will be defined as the percentage of participants in the intervention arm who are referred to and seen by supportive care services. The denominator will be all patients in the intervention arm who receive geriatric assessment-guided recommendations for supportive care referrals. The acceptability threshold will be met if ≥ 60% of these participants agree to and are seen by at least one recommended service during the study period. Will be summarized using descriptive statistics. Rates will be estimated along with the 95% exact binomial confidence interval. Analyses comparing groups of participants defined by response may be conducted by various two sample tests such as two-sample t-test or Wilcoxon rank sum test for the continuous endpoints, or Chi square test / Fisher's exact test for the categorical endpoints.
Proportion of any-grade non-hematologic treatment-related toxicities | Up to 3 months after completion of treatment
  Will be assessed in patients using CTCAE v 5.0. Will be summarized using descriptive statistics. For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Observed toxicities will be summarized by type, severity, and attribution. Rates will be estimated along with the 95% exact binomial confidence interval.
Patient/family caregiver self-reported outcomes | Up to 3 months after completion of treatment
  Will be assessed using the geriatric assessment, Functional Assessment of Cancer Therapy-Head and Neck questionnaire, distress thermometer, Montgomery Borgatta Caregiver Burden Scale, and satisfaction with communication. Will be summarized using descriptive statistics. For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Analyses comparing groups of participants defined by response may be conducted by various two sample tests such as two-sample t-test or Wilcoxon rank sum test for the continuous endpoints, or Chi square test / Fisher's exact test for the categorical endpoints.
Rate of unplanned readmissions | Up to 3 months after completion of treatment
  Will be summarized using descriptive statistics. Rates will be estimated along with the 95% exact binomial confidence interval. Analyses comparing groups of participants defined by response may be conducted by various two sample tests such as two-sample t-test or Wilcoxon rank sum test for the continuous endpoints, or Chi square test / Fisher's exact test for the categorical endpoints.
Rate of emergency room/urgent care visits | Up to 3 months after completion of treatment
  Will be summarized using descriptive statistics. Rates will be estimated along with the 95% exact binomial confidence interval. Analyses comparing groups of participants defined by response may be conducted by various two sample tests such as two-sample t-test or Wilcoxon rank sum test for the continuous endpoints, or Chi square test / Fisher's exact test for the categorical endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Arya Amini, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States